CLINICAL TRIAL: NCT02629848
Title: A Global Phase 3, Randomized, Placebo Controlled, Double-Blind Trial of AMG 706 in Combination With Paclitaxel and Carboplatin for Advanced Non-Squamous Non-Small Cell Lung Cancer (Asian Phase 3 Study)
Brief Title: Study of Motesanib (AMG 706) in Combination With Paclitaxel and Carboplatin for Advanced Non-Squamous Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to terminate the study because the study did not meet the primary endpoint.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TB-AB030103; U1111-1176-7347 (Registry Identifier: WHO); JapicCTI-121887 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Drug therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — motesanib diphosphate; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motesanib + Paclitaxel + Carboplatin (Experimental): Motesanib 125 mg, (5 x 25 mg) tablets, orally, once daily and paclitaxel 200 mg/m^2, intravenous, once on Day 1 and carboplatin at a dose to achieve a target Area Under the Curve (AUC) of 6.0 mg/mL x minute, once on Day 1 of a 3 week Cycle for up to 6 Cycles. After 6 Cycles, motesanib 125 mg, tablets, orally, once daily alone until disease progression, drug intolerability, study withdrawal or death for up to 36 months.
  Interventions: Drug: Motesanib; Drug: Paclitaxel; Drug: Carboplatin
- Placebo + Paclitaxel + Carboplatin (Placebo Comparator): Motesanib placebo-matching tablets, orally, once daily and paclitaxel 200 mg/m^2, intravenous, once on Day 1 and carboplatin at a dose to achieve a target AUC of 6.0 mg/mL x minute, once on Day 1 of a 3 week Cycle for up to 6 Cycles. After 6 Cycles, motesanib placebo-matching, tablets, orally, once daily alone until disease progression, drug intolerability, study withdrawal or death for up to 36 months.
  Interventions: Drug: Placebo; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Motesanib — Motesanib (AMG 706) 5 x 25 mg tablets
  Other Names: AMG 706
  Arms: Motesanib + Paclitaxel + Carboplatin
Drug: Placebo — Motesanib placebo-matching tablets
  Arms: Placebo + Paclitaxel + Carboplatin
Drug: Paclitaxel — Paclitaxel IV
Drug: Carboplatin — Carboplatin IV

SUMMARY:
This study will evaluate progression free survival (PFS), overall survival (OS), objective response rate (ORR), duration of response, and safety of motesanib (AMG706) in combination with paclitaxel and carboplatin compared to placebo in combination with paclitaxel and carboplatin.

DETAILED DESCRIPTION:
The drug being tested in this study is called motesanib. Motesanib is being tested in combination with paclitaxel and carboplatin to treat people who have Stage IV or recurrent non-squamous non-small cell lung cancer (NSCLC). This study will look at progression free survival, overall survival, overall response and safety.

The study enrolled 401 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which remained undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Motesanib 125 mg + Paclitaxel + Carboplatin
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient + Paclitaxel + Carboplatin

All participants were asked to take 5 X 25 mg motesanib tablets or placebo at the same time each day throughout the study. All participants received treatment with paclitaxel 200 mg/m^2 intravenous (IV) and carboplatin IV on Day 1 of each 3 week Cycle for up to 6 Cycles. After 6 Cycles participants could continue to receive motesanib or placebo alone for up to 36 months.

This multi-centre trial was conducted worldwide. The overall time to participate in this study was up to 36 months. Participants made multiple visits to the clinic, plus a final visit 30 days after receiving their last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

Disease Related:

1. Histologically or cytologically confirmed, Stage IV or recurrent non-squamous non-small cell lung cancer (NSCLC) (except diagnosis by sputum cytology only). Adenosquamous histology or an unclear histology subtype containing more than 10% squamous cells was not allowed.
2. No prior chemotherapy, molecularly-targeted therapy, or immunotherapy. Neoadjuvant and post-operative adjuvant therapy except chemotherapy with platinum agent completed 1 year prior to randomization was permitted.
3. Measurable or non-measurable lesion per Response Evaluation Criteria in Solid Tumor (RECIST) Version 1.1 criteria (except non-measurable lesion with malignant effusion only).
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
5. Life expectancy of ≥ 3 months as documented by the Investigator.

Demographic:

Must have been 18 years of age or older at the time informed consent was obtained.

Laboratory:

1. Hematological function, as follows:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L.
   * Platelet count ≥ 100 x 10^9/L and ≤ 850 x 10^9/L.
   * Hemoglobin ≥ 9 g/dL.
2. Renal function, as follows:

   * Creatinine clearance (GFR) > 40 mL/min (calculated by Cockcroft-Gault formula).
   * Urinary protein quantitative value of ≤ 30 mg in urinalysis or ≤ 1+ on dipstick unless total quantitative protein was < 500 mg in a 24-hour urine sample.
3. Hepatic function, as follows:

   * Aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN) or AST < 5 x ULN if liver metastases were present.
   * Alanine aminotransferase (ALT) ≤ 2.5 x ULN or ALT < 5 x ULN if liver metastases were present.
   * Alkaline phosphatase (ALP) ≤ 2.0 x ULN or ALP < 5 x ULN if liver or bone metastases were present.
   * Total bilirubin < 1.5 x ULN.
4. Coagulation function, as follows:

   * Partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1 x ULN.
   * International normalized ratio (INR) ≤ 1.5 x ULN.

Ethical:

Ability to give written informed consent.

General:

1. Able to take oral medications.
2. Able to start protocol-directed therapy within 7 days from the date of randomization.

Exclusion Criteria:

Disease Related:

1. Symptomatic central nervous system metastases. Participants with asymptomatic brain metastases were eligible if definitive therapy had been administered (surgery and/or radiation therapy), there was no planned treatment for brain metastasis, and the participant was clinically stable and off corticosteroids for at least 2 weeks prior to randomization. Participants with asymptomatic brain metastases were also eligible if the participant did not need definitive therapy (surgery and/or radiation therapy) or corticosteroids according to the Investigator's judgement.
2. Palliative radiation therapy:

   * Radiation therapy within 28 days prior to randomization for central (chest).
   * Radiation therapy within 14 days prior to randomization for distant metastatic foci.
3. History of pulmonary hemorrhage or gross hemoptysis (approximately 3 mL of bright red blood or more) within 6 months prior to randomization.

Medications:

1. Prior targeted therapies, including but not limited to:

   • AMG 706, inhibitors of vascular endothelial growth factor (VEGF) (eg, SU5416, SU6668, ZD6474, SU11248, PTK787, AZD2171, AEE-788, sorafenib, bevacizumab), or epidermal growth factor receptor (EGFR) (eg, panitumumab, cetuximab, gefitinib, erlotinib).
2. Any anticoagulation therapy within 7 days prior to randomization. The use of low-dose warfarin (≤ 2 mg daily) or low molecular weight heparin or heparin flushes for prophylaxis against central venous catheter thrombosis was allowed.
3. Known history of allergy or hypersensitivity reaction to paclitaxel or carboplatin.

General:

1. History of arterial or venous thrombosis within 12 months prior to randomization.
2. History of bleeding diathesis or bleeding within 14 days prior to randomization.
3. Peripheral neuropathy ≥ Grade 2 per Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0.
4. Clinically significant cardiovascular disease within 12 months of randomization, including myocardial infarction, unstable angina, ≥ Grade 2 peripheral vascular disease, cerebrovascular accident, transient ischemic attack, percutaneous transluminal coronary angioplasty/stent, congestive heart failure or ongoing arrhythmias requiring medication.
5. Any kind of disorder that compromised the ability of the participant to comply with the study procedures.
6. Open wound, ulcer or fracture.
7. Active or any uncontrolled, infection or inflammatory disease requiring systemic treatment ≤ 14 days prior to randomization.
8. Diagnosed interstitial lung disease and/or significant interstitial shadow on the computerized tomography (CT) image.
9. Uncontrolled hypertension as defined by resting blood pressure > 150/90 mmHg despite the use of an antihypertensive.
10. History (past/current) of other primary cancer unless:

    * Curatively resected non-melanomatous skin cancer.
    * Curatively treated cervical carcinoma in situ.
    * Other primary solid tumor curatively treated with no known active disease present and no curative treatment administered for the last 3 years.
11. Surgery:

    * Major surgical procedures within 28 days prior to randomization.
    * Minor surgical procedures within 14 days prior to randomization.
    * Failure to recover from prior surgery.
    * Placement of a central venous access device (including ports and tunneled or non-tunneled catheters) within 3 days in principle prior to randomization.
    * Core needle biopsy within 7 days prior to randomization.
12. Planned elective surgery while on the study treatment.
13. Not recovered from all previous therapies (ie, radiation, surgery and medications). AEs related to previous therapies must have been CTCAE Grade ≤ 1 at Screening or must have resolved to the participant's Baseline level prior to the most recent previous therapy (except alopecia).
14. Participation in therapeutic clinical trials or currently receiving other investigational treatment(s) within 30 days prior to randomization.
15. Pregnant (eg, positive human chorionic gonadotropin [HCG] test-urine or serum) or breast-feeding woman.
16. Any participant not consenting to use adequate contraceptive precautions, from informed consent until 6 months after the last treatment.
17. Known to be human immunodeficiency virus (HIV), hepatitis B surface (HBs) antigen or hepatitis C positive. Participants may have been HBs antigen (-) and HB core antibody (+) and /or HBs antibody (+) with hepatitis B virus (HBV) deoxyribonucleic acid (DNA) (-). If HBs antigen (-) but HBV DNA (+), participant could be enrolled with concomitant antiviral treatment (entecavir or tenofovir). In case of hepatitis C virus (HCV) antibody (+) with HCV ribonucleic acid (-) and/or HCV core antigen (-), participants could be enrolled.

    Participant with HBs antigen (+) could be enrolled if AST and ALT were within ULN, and HBV DNA level was less than 3.0 Log. The participant must have received concomitant antiviral treatment (entecavir or tenofovir). Participants who were already on antiviral treatment at Screening were not eligible.
18. Known chronic hepatitis.
19. History of any medical or psychiatric condition or laboratory abnormality that, in the opinion of the Investigator, may have increased the risks associated with participation in the study or administration of investigational products (IPs) administration, or may have interfered with the interpretation of the results.
20. Previously randomized to this study.
21. Not available for follow-up assessments or unable to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Up to 24 Months
  PFS was defined as the time from the date of randomization to the date of disease progression per Response Evaluation Criteria in Solid Tumor (RECIST) Version 1.1 or death from any cause, whichever occurred first. Progressive disease was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.

SECONDARY OUTCOMES:
Overall Survival (OS) | 6, 12, 18 and 24 months
  OS was defined as the time from randomization to death (or, where applicable, the censoring date). Participants who had not died or were lost to follow-up by the analysis data cut-off date were censored at their last contact date. Participants who withdrew full consent to participate in the study were censored on the date consent was withdrawn.
Objective Response Rate (ORR) | Up to 30 months
  ORR was defined as the percentage of participants achieving either a complete response (CR) or partial response (PR) per RECIST Version 1.1 criteria. CR= disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. PR= At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the Baseline sum LD.
Duration of Response (DOR) | Up to 30 months
  DOR was defined as the time from the date of first response (CR or PR) to disease progression (per RECIST Version 1.1) or death. CR= Disappearance of all target lesions; disappearance of all non-target lesions and normalization of tumor marker level. PR= At least a 30% decrease in the sum of the longest diameter (LD ) of target lesions, taking as reference the Baseline sum LD.
Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to 30 months
  An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Percentage of Participants with Abnormal Clinical Laboratory Findings | Up to 30 months
  The percentage of participants with any chemistry or hematology abnormal standard safety laboratory values collected throughout study
Cmax: Maximum Observed Plasma Concentration for Montesanib and its Metabolite M4 | Predose on Day 1 and 1 to 2 hours postdose in Cycles 3 and 5
  Maximum Observed Plasma Concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration- time curve.
Cmin: Minimum Observed Plasma Concentration for Montesanib and its Metabolite M4 | Predose on Day 1 and 1 to 2 hours postdose in Cycles 3 and 5
  Minimum observed plasma concentration (Cmin) is the lowest plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda